CLINICAL TRIAL: NCT03100942
Title: A Randomized, Phase 2, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of Filgotinib, GS-9876 and GS-4059 in Adult Subjects With Active Sjogren's Syndrome
Brief Title: Study to Assess Safety and Efficacy of Filgotinib, Lanraplenib and Tirabrutinib in Adults With Active Sjogren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry); Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-445-4189; 2016-003558-34 (EudraCT Number)
Record Dates: First submitted 2017-03-31; First posted 2017-04-04 (Actual); Results first posted 2020-01-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — GLPG0634; tirabrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lanraplenib (Experimental): Lanraplenib + filgotinib placebo + tirabrutinib placebo for up to 49.4 weeks.
  Interventions: Drug: Lanraplenib; Drug: Filgotinib placebo; Drug: Tirabrutinib placebo
- Filgotinib (Experimental): Filgotinib + lanraplenib placebo + tirabrutinib placebo for up to 50.4 weeks.
  Interventions: Drug: Filgotinib; Drug: Lanraplenib placebo; Drug: Tirabrutinib placebo
- Tirabrutinib (Experimental): Tirabrutinib + filgotinib placebo + lanraplenib placebo for up to 50.3 weeks.
  Interventions: Drug: Tirabrutinib; Drug: Lanraplenib placebo; Drug: Filgotinib placebo
- Placebo, then active treatment (Placebo Comparator): Filgotinib placebo + lanraplenib placebo + tirabrutinib placebo for 24 weeks. Following completion of the Week 24 assessments and procedures, participants will be rerandomized 1:1:1, in a blinded fashion and receive either of the following study drugs through Week 48:
  * filgotinib + lanraplenib placebo + tirabrutinib placebo
  * lanraplenib + filgotinib placebo + tirabrutinib placebo
  * tirabrutinib + filgotinib placebo + lanraplenib placebo
  Interventions: Drug: Lanraplenib; Drug: Filgotinib; Drug: Tirabrutinib; Drug: Lanraplenib placebo; Drug: Filgotinib placebo; Drug: Tirabrutinib placebo

INTERVENTIONS:
Drug: Lanraplenib — 1 x 30 mg tablet administered orally once daily
  Other Names: GS-9876
  Arms: Lanraplenib; Placebo, then active treatment
Drug: Filgotinib — 1 x 200 mg tablet administered orally once daily
  Other Names: GS-6034
  Arms: Filgotinib; Placebo, then active treatment
Drug: Tirabrutinib — 1 x 40 mg tablet administered orally once daily
  Other Names: GS-4059
  Arms: Placebo, then active treatment; Tirabrutinib
Drug: Lanraplenib placebo — 1 x tablet administered orally once daily
  Arms: Filgotinib; Placebo, then active treatment; Tirabrutinib
Drug: Filgotinib placebo — 1 x tablet administered orally once daily
  Arms: Lanraplenib; Placebo, then active treatment; Tirabrutinib
Drug: Tirabrutinib placebo — 1 x tablet administered orally once daily
  Arms: Filgotinib; Lanraplenib; Placebo, then active treatment

SUMMARY:
The primary objective of this study is to assess the efficacy of filgotinib, lanraplenib, and tirabrutinib in adults with active Sjogren's Syndrome (SjS).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with primary or secondary SjS according to the 2002 American European Consensus Group (AECG) classification
* Active SjS as defined by an European League Against Rheumatism (EULAR) Sjogren's syndrome disease activity index (ESSDAI) ≥ 5
* Seropositivity for antibodies to SjS-associated antigens A and/or B (anti-SSA or anti-SSB)

Key Exclusion Criteria:

* Concurrent treatment with any biologic disease modifying antirheumatic drug (bDMARD) (prior bDMARD treatment allowed with appropriate washout as per study protocol)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (53):
- United States (34):
  - AARR Arizona Arthritis & Rheumatology Research, Mesa, Arizona
  - AARR Arizona Arthritis & Rheumatology Research, Phoenix, Arizona
  - Medvin Clinical Research, Covina, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Omega Research Consultants LLC, DeBary, Florida
  - Center for Rheumatology Immunology and Arthritis, Fort Lauderdale, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - IRIS Research and Development, LLC, Plantation, Florida
  - North Georgia Rheumatology Group, PC, Lawrenceville, Georgia
  - Springfield Clinic, Springfield, Illinois
  - Center for Arthritis & Osteoporosis, Elizabethtown, Kentucky
  - June DO, PC, Lansing, Michigan
  - North Mississippi Medical Clinics, Inc. - Clinical Research, Tupelo, Mississippi
  - Clayton Medical Associates, St Louis, Missouri
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - Cape Fear Arthritis Care, PLLC, Leland, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - East Penn Rheumatology Associates, P.C., Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - ClinSearch, Chattanooga, Tennessee
  - Ramesh C. Gupta, MD, Memphis, Tennessee
  - Diagnostic Group Integrated Healthcare System, Pllc, Beaumont, Texas
  - Accurate Clinical Research Inc., Houston, Texas
  - Southwest Rheumatology Research, Mesquite, Texas
  - Trinity Universal Research Associates, Plano, Texas
  - Arthritis & Osteoporosis Clinic, Waco, Texas
  - Wasatch Peak Family Practice, Layton, Utah
  - The Center for Arthritis and Rheumatic Diseases, PC, Chesapeake, Virginia
  - Arthritis Northwest, Spokane, Washington
- Poland (6):
  - Centrum Kliniczno-Badawcze, Elblag
  - Intermedius, Kościan
  - Centrum Badan Klinicznych S.C, Poznan
  - Ai Centrum Medyczne, Poznan
  - Centrum Medyczne Amed Warszawa Targowek, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
- Spain (8):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario De Elche, Elche
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital De Merida, Mérida
  - Corporacio Sanitaria Parc Taulí de Sabadell, Sabadell
  - Hospital Clinico Universitario de Salamanca, San Vicente
  - Hospital Quironsalud Infanta Luisa, Seville
- United Kingdom (5):
  - Doncaster Royal Infirmary, Doncaster
  - Western General Hospital, Edinburgh
  - Princess Alexandra Hospital, Harlow
  - Great Western Hospital, Swindon
  - Warrington Hospital, Warrington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Price E, Bombardieri M, Kivitz A, Matzkies F, Gurtovaya O, Pechonkina A, Jiang W, Downie B, Mathur A, Mozaffarian A, Mozaffarian N, Gottenberg JE. Safety and efficacy of filgotinib, lanraplenib and tirabrutinib in Sjogren's syndrome: a randomized, phase 2, double-blind, placebo-controlled study. Rheumatology (Oxford). 2022 Nov 28;61(12):4797-4808. doi: 10.1093/rheumatology/keac167. PMID 35377447

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and Europe. The first participant was screened on 01 May 2017. The last study visit occurred on 02 October 2019.
Pre-assignment Details: 348 participants were screened.
Groups:
- Lanraplenib: Lanraplenib (1 x 30 mg tablet) + filgotinib placebo (1 x tablet) + tirabrutinib placebo (1 x tablet) orally once daily for up to 49.4 weeks.
- Filgotinib: Filgotinib (1 x 200 mg tablet) + lanraplenib placebo (1 x tablet) + tirabrutinib placebo (1 x tablet) orally once daily for up to 50.4 weeks
- Tirabrutinib: Tirabrutinib (1 x 40 mg tablet) + filgotinib placebo (1 x tablet) + lanraplenib placebo (1 x tablet) orally once daily for up to 50.3 weeks
- Placebo: Participants received filgotinib placebo + lanraplenib placebo + tirabrutinib placebo tablets orally once daily for 24 weeks.
  At Week 24 visit, participants were re-randomized 1:1:1, in a blinded fashion and receive either of the following study drugs through Week 48:
  * filgotinib + lanraplenib placebo + tirabrutinib placebo
  * lanraplenib + filgotinib placebo + tirabrutinib placebo
  * tirabrutinib + filgotinib placebo + lanraplenib placebo
- Placebo to Lanraplenib: Participants who received placebo for 24 weeks were re-randomized at the Week 24 visit and received lanraplenib (1 × 30 mg tablet) + filgotinib placebo (1 × tablet) + tirabrutinib placebo (1 × tablet) orally once daily for up to 25.1 weeks.
- Placebo to Filgotinib: Participants who received placebo for 24 weeks were re-randomized at the Week 24 visit and received filgotinib (1 × 200 mg tablet) + lanraplenib placebo (1 × tablet) + tirabrutinib placebo (1 × tablet) orally once daily for up to 24.4 weeks.
- Placebo to Tirabrutinib: Participants who received placebo for 24 weeks were re-randomized at the Week 24 visit and received tirabrutinib (1 × 40 mg tablet) + filgotinib placebo (1 × tablet) + lanraplenib placebo (1 × tablet) orally once daily for up to 24.9 weeks.
Period: Randomized Treatment Period
Arm/Group | Lanraplenib | Filgotinib | Tirabrutinib | Placebo | Placebo to Lanraplenib | Placebo to Filgotinib | Placebo to Tirabrutinib
Started | 38 | 38 | 39 | 37 | 0 | 0 | 0
Completed | 26 | 29 | 33 | 32 | 0 | 0 | 0
Not Completed | 12 | 9 | 6 | 5 | 0 | 0 | 0
Not completed — Withdrew Consent | 4 | 5 | 3 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Investigator's Discretion | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Randomized but Didn't Receive Study Drug | 1 | 0 | 0 | 1 | 0 | 0 | 0
Period: Placebo Arm Re-Randomized
Arm/Group | Lanraplenib | Filgotinib | Tirabrutinib | Placebo | Placebo to Lanraplenib | Placebo to Filgotinib | Placebo to Tirabrutinib
Started | 0 | 0 | 0 | 0 | 10 | 12 | 10
Completed | 0 | 0 | 0 | 0 | 10 | 12 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received filgotinib placebo + lanraplenib placebo + tirabrutinib placebo tablets orally once daily for 24 weeks. At Week 24 Visit, participants were rerandomized 1:1:1, in a blinded fashion and received either of the three experimental study drugs orally once daily through Week 48:
  * lanraplenib (1 x 30 mg tablet) + filgotinib placebo (1 x tablet) + tirabrutinib placebo (1 x tablet)
  * filgotinib (1 x 200 mg tablet) + lanraplenib placebo (1 x tablet) + tirabrutinib placebo (1 x tablet)
  * tirabrutinib (1 x 40 mg tablet) + filgotinib placebo (1 x tablet) + lanraplenib placebo (1 x tablet)
- Total: Total of all reporting groups
Arm/Group | Lanraplenib | Filgotinib | Tirabrutinib | Placebo | Total
Number analyzed (Participants) | 37 | 38 | 39 | 36 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (9.72) | 52.2 (10.54) | 55.8 (10.06) | 53.2 (10.28) | 54.4 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 37 | 35 | 146
  Male | 1 | 0 | 2 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 1 | 6 | 17
  Not Hispanic or Latino | 31 | 34 | 38 | 30 | 133
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 1 | 0 | 2
  Black | 5 | 5 | 4 | 5 | 19
  White | 31 | 32 | 34 | 30 | 127
  Other | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 30 | 23 | 106
  Poland | 7 | 4 | 5 | 6 | 22
  Spain | 2 | 4 | 3 | 4 | 13
  United Kingdom | 2 | 3 | 1 | 3 | 9
European League Against Rheumatism (EULAR) Sjogren's syndrome disease activity index (ESSDAI) [Mean (Standard Deviation); unit: Score on a scale] — Overall score (ranged from 0 (best) to 123 (worst activity)) was calculated as sum of all individual weighted domain scores. For additional details on this index, please see Outcome Measures# 2 and 4.
  Score on a scale | 10.5 (4.89) | 10.2 (6.23) | 10.4 (5.36) | 9.3 (3.96) | 10.1 (5.16)
EULAR Sjogren's syndrome patient reported index (ESSPRI) [Mean (Standard Deviation); unit: Score on a scale] — The ESSPRI is a patient-reported questionnaire to assess subjective patient symptoms and includes 3 domains (dryness, pain, and fatigue). Each domain scored on scale of 0-10 (0 = no symptoms at all and 10 = worst symptoms imaginable), and an overall score is calculated as the mean of the three individual domain scores where all domains carry the same weight. Minimum score can be 0 and maximum score can be 10.
  Score on a scale | 6.6 (1.90) | 6.3 (2.31) | 5.9 (2.39) | 5.9 (2.24) | 6.2 (2.22)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Fulfilling Protocol-Specified Response Criteria at Week 12, as Compared to Baseline
Description: Response was defined as: Improvement ≥ 20% in ≥ 3 of 5 participant-reported Sjogren's syndrome (SjS) related visual analogue score (VAS) measures (participant's assessment of global disease, pain, oral dryness, ocular dryness and fatigue), with no increase defined as > 30 mm from baseline (Day 1) in any of the above 5 VAS measures, AND either ≥ 20% improvement in high sensitivity C-reactive protein (hsCRP) (if hsCRP ≥ 1.5 x upper limit of normal [ULN] on Day 1) or no increase in hsCRP to ≥ 1.5 x ULN (if hsCRP < 1.5 x ULN on Day 1).
Time Frame: Week 12
Population: The Full Analysis Set included all randomized participants who received at least one dose of study drug. Included participants with available data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Lanraplenib: Lanraplenib (1 x 30 mg tablet) + filgotinib placebo (1 x tablet) + tirabrutinib placebo (1 x tablet) orally once daily for 48 weeks
- Filgotinib: Filgotinib (1 x 200 mg tablet) + lanraplenib placebo (1 x tablet) + tirabrutinib placebo (1 x tablet) orally once daily for 48 weeks
- Tirabrutinib: Tirabrutinib (1 x 40 mg tablet) + filgotinib placebo (1 x tablet) + lanraplenib placebo (1 x tablet) orally once daily for 48 weeks
- Placebo: Participants received filgotinib placebo + lanraplenib placebo + tirabrutinib placebo tablets orally once daily for 24 weeks. At Week 24 Visit, participants were rerandomized 1:1:1, in a blinded fashion and received either of the three experimental study drugs orally once daily through Week 48:
  * filgotinib (1 x 200 mg tablet) + lanraplenib placebo (1 x tablet) + tirabrutinib placebo (1 x tablet)
  * lanraplenib (1 x 30 mg tablet) + filgotinib placebo (1 x tablet) + tirabrutinib placebo (1 x tablet)
  * tirabrutinib (1 x 40 mg tablet) + filgotinib placebo (1 x tablet) + lanraplenib placebo (1 x tablet)
Arm/Group | Lanraplenib | Filgotinib | Tirabrutinib | Placebo
Number analyzed (Participants) | 35 | 37 | 37 | 34
percentage of participants | 42.9 [25.0 to 60.7] | 43.2 [25.9 to 60.6] | 35.1 [18.4 to 51.9] | 26.5 [10.2 to 42.8]
Statistical Analysis 1: Comparison: Lanraplenib vs Placebo; Test type: Superiority; p = 0.1597, Cochran-Mantel-Haenszel — P-values were obtained from Cochran-Mantel-Haenszel (CMH) test stratified by randomization stratification factors; Difference in Response Rates = 15.6, 95% CI 2-sided [-6.3 to 37.6] — For the analysis of the difference in response rates, the data with missing response values were imputed by multiple imputation method with logistic regression
Statistical Analysis 2: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.1694, Cochran-Mantel-Haenszel — P-values were obtained from CMH test stratified by randomization stratification factors; Difference in Response Rates = 16.6, 95% CI 2-sided [-5.1 to 38.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Tirabrutinib vs Placebo; Test type: Superiority; p = 0.3309, Cochran-Mantel-Haenszel — P-values were obtained from CMH test stratified by randomization stratification factors; Difference in Response Rates = 8.1, 95% CI 2-sided [-13.2 to 29.4] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in European League Against Rheumatism (EULAR) Sjogren's Syndrome Disease Activity Index (ESSDAI) at Week 12
Description: The ESSDAI is a physician-administered tool designed to measure disease activity. It consists of 12 organ-specific 'domains' contributing to disease activity associated with the participant's Sjogren's Syndrome only (constitutional, lymphadenopathy, articular, muscular, cutaneous, glandular, pulmonary, renal, peripheral nervous system, central nervous system, hematological, biological). Each domain is assessed for activity level (i.e., no, low, moderate, high) and assigned a numerical score based on pre-determined weighting of each individual domain. Overall score (ranges from 0 (no activity) to 123 (worst activity)) is calculated as sum of all individual weighted domain scores. A negative change from baseline value indicates improvement.
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lanraplenib | Filgotinib | Tirabrutinib | Placebo
Number analyzed (Participants) | 37 | 38 | 39 | 36
score on a scale | -2.5 (0.76) | -4.7 (0.72) | -3.2 (0.73) | -3.9 (0.76)
Statistical Analysis 1: Comparison: Lanraplenib vs Placebo; Least Squares (LS) Means, 95% confidence interval (CI), and P-values were obtained from Mixed Effects Model for Repeated Measures (MMRM) with the terms for baseline value, treatment, stratification factors, visit, and treatment-by-visit interaction; Test type: Superiority; p = 0.2066, MMRM; LS Mean Difference = 1.3, 95% CI 2-sided [-0.7 to 3.4], Standard Error of Mean 1.05
Statistical Analysis 2: Comparison: Filgotinib vs Placebo; LS Means, 95% CI, and P-values were obtained from MMRM with the terms for baseline value, treatment, stratification factors, visit, and treatment-by-visit interaction; Test type: Superiority; p = 0.3998, MMRM; LS Mean Difference = -0.9, 95% CI 2-sided [-2.9 to 1.2], Standard Error of Mean 1.04
Statistical Analysis 3: Comparison: Tirabrutinib vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.5113, MMRM; LS Mean Difference = 0.7, 95% CI 2-sided [-1.4 to 2.7], Standard Error of Mean 1.04

3. Secondary Outcome: Change From Baseline in EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) at Week 12
Description: The ESSPRI is a participant-reported questionnaire to assess subjective participant symptoms and includes 3 domains (dryness, pain, and fatigue). Each domain is scored on scale of 0-10 (0 = no symptom at all and 10 = worst symptom imaginable), and an overall score is calculated as the mean of the three individual domains where all domains carry the same weight. Minimum score can be 0 and maximum score can be 10. A negative change from baseline value indicates improvement.
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lanraplenib | Filgotinib | Tirabrutinib | Placebo
Number analyzed (Participants) | 37 | 38 | 39 | 36
score on a scale | -1.0 (0.34) | -1.4 (0.33) | -1.4 (0.33) | -1.0 (0.34)
Statistical Analysis 1: Comparison: Lanraplenib vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.9446, MMRM; LS Mean Difference = 0.0, 95% CI 2-sided [-0.9 to 1.0], Standard Error of Mean 0.47
Statistical Analysis 2: Comparison: Filgotinib vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.3977, MMRM; LS Mean Difference = -0.4, 95% CI 2-sided [-1.3 to 0.5], Standard Error of Mean 0.47
Statistical Analysis 3: Comparison: Tirabrutinib vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.4966, MMRM; LS Mean Difference = -0.3, 95% CI 2-sided [-1.2 to 0.6], Standard Error of Mean 0.47

4. Secondary Outcome: Change From Baseline in ESSDAI at Week 24
Description: as for outcome 2
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lanraplenib | Filgotinib | Tirabrutinib | Placebo
Number analyzed (Participants) | 37 | 38 | 39 | 36
score on a scale | -4.3 (0.81) | -5.4 (0.75) | -4.0 (0.75) | -4.2 (0.78)
Statistical Analysis 1: Comparison: Lanraplenib vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.9564, MMRM; LS Mean Difference = -0.1, 95% CI 2-sided [-2.2 to 2.1], Standard Error of Mean 1.10
Statistical Analysis 2: Comparison: Filgotinib vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.2788, MMRM; LS Mean Difference = -1.2, 95% CI 2-sided [-3.3 to 0.9], Standard Error of Mean 1.07
Statistical Analysis 3: Comparison: Tirabrutinib vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.8047, MMRM; LS Mean Difference = 0.3, 95% CI 2-sided [-1.8 to 2.3], Standard Error of Mean 1.06

5. Secondary Outcome: Change From Baseline in ESSPRI at Week 24
Description: as for outcome 3
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lanraplenib | Filgotinib | Tirabrutinib | Placebo
Number analyzed (Participants) | 37 | 38 | 39 | 36
score on a scale | -1.1 (0.34) | -0.8 (0.31) | -1.2 (0.31) | -0.9 (0.33)
Statistical Analysis 1: Comparison: Lanraplenib vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.6782, MMRM; LS Mean Difference = -0.2, 95% CI 2-sided [-1.1 to 0.7], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: Filgotinib vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.9171, MMRM; LS Mean Difference = 0.0, 95% CI 2-sided [-0.8 to 0.9], Standard Error of Mean 0.45
Statistical Analysis 3: Comparison: Tirabrutinib vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.4641, MMRM; LS Mean Difference = -0.3, 95% CI 2-sided [-1.2 to 0.5], Standard Error of Mean 0.45

ADVERSE EVENTS:
Time Frame: First dose date up to last dose date (Maximum: 50.4 weeks) plus 30 days
Description: The Safety Analysis Set included participants who received at least one dose of study drug.
Groups:
- Placebo to Lanraplenib: Participants who received placebo for 24 weeks were rerandomized at the Week 24 visit and received lanraplenib (1 × 30 mg tablet) + filgotinib placebo (1 × tablet) + tirabrutinib placebo (1 × tablet) orally once daily for up to 25.1 weeks.
- Placebo to Filgotinib: Participants who received placebo for 24 weeks were rerandomized at the Week 24 visit and received filgotinib (1 × 200 mg tablet) + lanraplenib placebo (1 × tablet) + tirabrutinib placebo (1 × tablet) orally once daily for up to 24.4 weeks.
- Placebo to Tirabrutinib: Participants who received placebo for 24 weeks were rerandomized at the Week 24 visit and received tirabrutinib (1 × 40 mg tablet) + filgotinib placebo (1 × tablet) + lanraplenib placebo (1 × tablet) orally once daily for up to 24.9 weeks.
- Placebo on Placebo Controlled Period: Participants received filgotinib placebo + lanraplenib placebo + tirabrutinib placebo tablets orally once daily for 24 weeks in placebo controlled period.
  At Week 24 visit, participants were re-randomized 1:1:1, in a blinded fashion and receive either of the following study drugs through Week 48:
  * filgotinib + lanraplenib placebo + tirabrutinib placebo
  * lanraplenib + filgotinib placebo + tirabrutinib placebo
  * tirabrutinib + filgotinib placebo + lanraplenib placeboy once daily for 24 weeks.
Arm/Group | Lanraplenib | Filgotinib | Tirabrutinib | Placebo to Lanraplenib | Placebo to Filgotinib | Placebo to Tirabrutinib | Placebo on Placebo Controlled Period
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38 | 0/39 | 0/10 | 0/12 | 0/10 | 0/36
Serious Adverse Events (participants affected / at risk) | 3/37 | 5/38 | 1/39 | 0/10 | 1/12 | 0/10 | 2/36
Other Adverse Events (participants affected / at risk) | 30/37 | 31/38 | 32/39 | 10/10 | 10/12 | 7/10 | 23/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lanraplenib (N=37) | Filgotinib (N=38) | Tirabrutinib (N=39) | Placebo to Lanraplenib (N=10) | Placebo to Filgotinib (N=12) | Placebo to Tirabrutinib (N=10) | Placebo on Placebo Controlled Period (N=36)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lanraplenib (N=37) | Filgotinib (N=38) | Tirabrutinib (N=39) | Placebo to Lanraplenib (N=10) | Placebo to Filgotinib (N=12) | Placebo to Tirabrutinib (N=10) | Placebo on Placebo Controlled Period (N=36)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 0
Corneal erosion (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 3 | 1 | 2 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Lip blister (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 2 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 2 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 4 | 0 | 3 | 2 | 1 | 0 | 2
Pyrexia (General disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 1 | 2 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 3 | 1 | 0 | 1 | 0 | 3
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 3 | 2 | 3 | 2 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 3 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 6 | 4 | 1 | 1 | 2 | 4
Oral herpes (Infections and infestations) | 2 | 3 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 5 | 1 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 9 | 0 | 1 | 0 | 4
Urinary tract infection (Infections and infestations) | 1 | 2 | 4 | 2 | 2 | 0 | 6
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 2 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Light chain analysis increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 6 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 3 | 3 | 1 | 1 | 1 | 1
Migraine (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 0 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 3 | 0 | 0 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 3 | 0 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
An unplanned review of unblinded clinical trial data was performed in this study that was not prospectively specified in the protocol. There was no impact on the overall integrity or conclusions of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03100942/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT03100942/SAP_001.pdf